CLINICAL TRIAL: NCT06102824
Title: Organoid-Guided Functional Precision Therapy Versus Treatment of Physician's Choice in Previously Treated HER2-negative Advanced Breast Cancer: A Phase II, Multicenter, Open-label, Randomized Controlled Trial
Brief Title: Organoid-based Functional Precision Therapy for Advanced Breast Cancer
Acronym: ORIENTA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-sen University (Other); Shantou Central Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, M.D., Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20231028
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: HER2-negative Breast Cancer; Advanced Breast Cancer
Keywords: HER2-negative; Advanced breast cancer; Patient-derived organoids; Precision medicine; Randomized
MeSH Terms: interventions — taxane; Albumin-Bound Paclitaxel; Capecitabine; Gemcitabine; Vinorelbine; eribulin; Anthracyclines; liposomal doxorubicin; Carboplatin; trastuzumab deruxtecan; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Organoid-guided treatment (Experimental): Subjects randomized to the organoid-guided treatment (OGT) group will be treated with the drugs predicted to be the most sensitive through PDO drug sensitivity screening. Drugs that the subjects have progressed on before randomization will not be screened. The drugs selected for organoid screening are from the following options: taxane, anthracycline, 5-fluorouracil, gemcitabine, vinorelbine, eribulin, utidelone, carboplatin, sacituzumab govitecan, and trastuzumab deruxtecan (for HER2-low patients).
  Interventions: Drug: Organoid-guided treatment
- Treatment of physician's choice (Active Comparator): Subjects randomized to the treatment of physician's choice (TPC) group will receive physician-chosen therapy from the following options: taxane, anthracycline, 5-fluorouracil, gemcitabine, vinorelbine, eribulin, utidelone, carboplatin, sacituzumab govitecan, and trastuzumab deruxtecan (for HER2-low patients).
  Interventions: Drug: Taxane; Drug: Capecitabine; Drug: Gemcitabine; Drug: Vinorelbine; Drug: Eribulin; Drug: Anthracycline; Drug: Carboplatin; Drug: Utidelone; Drug: Trastuzumab deruxtecan; Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Organoid-guided treatment — The drugs predicted to be the most sensitive through organoid drug sensitivity screening. The drugs selected for sensitivity screening are from the following options: taxane, anthracycline, 5-fluorouracil, gemcitabine, vinorelbine, eribulin, utidelone, carboplatin, sacituzumab govitecan, and trastuzumab deruxtecan (for HER2-low patients).
  Arms: Organoid-guided treatment
Drug: Taxane — Albumin-bound paclitaxel 260mg/m2, IV, q3w, or 100-125mg/m2, IV, days 1, 8, and 15, q4w OR Liposomal paclitaxel 175mg/m2, IV, q3w
  Other Names: Abraxane, Lipusu
  Arms: Treatment of physician's choice
Drug: Capecitabine — 1000-1250mg/m2, PO, bid, days1-14, q3w
  Other Names: Xeloda
  Arms: Treatment of physician's choice
Drug: Gemcitabine — 800-1200mg/m2, IV, days 1, 8, q3w
  Other Names: Gemzar
  Arms: Treatment of physician's choice
Drug: Vinorelbine — 20-35mg/m2, IV, days 1 and 8, q3w
  Other Names: Navelbine
  Arms: Treatment of physician's choice
Drug: Eribulin — 1.4mg/m2, IV, days 1 and 8, q3w
  Other Names: Halaven
  Arms: Treatment of physician's choice
Drug: Anthracycline — Liposomal doxorubicin 50mg/m2, IV, q3w OR Liposomal doxorubicin 40mg/m2+Cyclophosphamide 600mg/m2, IV, q3w
  Other Names: Doxil, Lipodox
  Arms: Treatment of physician's choice
Drug: Carboplatin — Carboplatin AUC 6, IV, q3w or q4w OR Carboplatin AUC 2+Gemcitabine 1000mg/m2, IV, days 1 and 8, q3w OR Carboplatin AUC 2+Albumin-bound paclitaxel 125mg/m2, IV, days 1 and 8, q3w
  Other Names: Paraplatin
  Arms: Treatment of physician's choice
Drug: Utidelone — 30mg/m2, IV, once per day on days 1-5, q3w
  Other Names: UTD1
  Arms: Treatment of physician's choice
Drug: Trastuzumab deruxtecan — 5.4mg/kg, IV, q3w
  Other Names: Enhertu
  Arms: Treatment of physician's choice
Drug: Sacituzumab govitecan — 10mg/kg, IV, days 1 and 8, q3w
  Other Names: Trodelvy
  Arms: Treatment of physician's choice

SUMMARY:
This is a phase II, multicenter, open-label, randomized controlled trial to compare the efficacy of organoid-guided treatment (OGT) to treatment of physician's choice (TPC) in previously treated, HER2-negative locally advanced or metastatic breast cancer. The study will seek to provide evidence for utilizing patient-derived organoid (PDO) model to personalize treatment strategies and inform clinical care for advanced breast cancer. Subjects randomized to the OGT group will undergo PDO generation and receive treatment dictated by subsequent PDO drug sensitivity screening. Subjects randomized to the TPC group will receive empirical therapy as selected by the treating physician.

DETAILED DESCRIPTION:
Treatment for advanced-stage breast cancer has long been challenging. Genomic-based precision medicine was able to facilitate treatment selection in some patients, but there were considerable instances where genomic profiling failed to assign effective interventions or patients exhibited refractoriness to the drugs nominated by genomic alterations. Patient-derived organoids (PDOs) represent a tractable tool that may compensate for the drawbacks of genomic medicine to identify therapeutic opportunities in rare or metastatic cancers. Previous research has demonstrated that PDOs displayed strong biological fidelity to their original tumors and functional precision medicine based on PDO drug screening could confer survival benefits in breast cancer patients.

This multicenter, open-label, randomized phase II trial aims to investigate the safety and efficacy of organoid-guided treatment (OGT) versus treatment of physician's choice (TPC) in previously treated, HER2-negative locally advanced or metastatic breast cancer. Randomization will be stratified by hormone receptor status and prior chemotherapy for the advanced or metastatic disease. Subjects in the OGT group will receive treatment predicted to be the most efficacious by the PDO drug sensitivity screening, and subjects in the TPC group will receive treatment selected by the treating physician. Treatments tested in PDO drug screening or chosen by the treating physician will be guided by NCCN guidelines. Treatment that subjects have previously received before randomization is no longer subjected to PDO sensitivity screening. This study will provide valuable evidence on the real-time application of PDOs in the context of clinical care.

ELIGIBILITY:
Inclusion Criteria:

1. Must be competent and able to comprehend, sign, and date a written informed consent form (ICF) before performance of any study-specific procedures or tests.
2. Men or women ≥18 years old.
3. Pathologically documented unresectable locally advanced or metastatic breast cancer that:

   3.1 Confirmed as HER2-negative status, defined as IHC 0, IHC 1+, or IHC 2+/ISH- according to American Society of Clinical Oncology College of American Pathologists (ASCO/CAP) guidelines evaluated at a local laboratory.

   3.2 Is HR-positive or HR-negative. Positive for estrogen receptor or progesterone receptor if a finding of ≥1% of tumor cell nuclei is immunoreactive according to ASCO/CAP guidelines.

   3.3 Has been treated with at least 1 prior line of systemic therapy in the advanced or metastatic setting. If >10% ER expression, the subject should have been treated with a CDK4/6 inhibitor. If recurrence occurred within 6 months of adjuvant chemotherapy, adjuvant therapy would count as 1 line of systemic therapy. If recurrence occurred within 12 months of adjuvant CDK4/6 inhibitor and endocrine therapy, adjuvant therapy would count as 1 line of systemic therapy.
4. Documented radiologic progression (during or after most recent treatment).
5. Presence of at least 1 measurable lesion based on computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
7. All subjects must have a recent tumor sample after the most recent treatment regimen or agree to undergo a tissue biopsy prior to randomization.
8. No visceral crisis.
9. Life expectancy of ≥ 6 months as assessed by the treating investigator.
10. Complete all required baseline laboratory tests and imaging examinations within 28 days before randomization.
11. Normal organ and bone marrow function measured within 28 days prior to administration of study treatment.
12. Male and female subjects of reproductive/childbearing potential must have a documented negative pregnancy test within 2 weeks prior to randomization and agree to acceptable birth control (non-hormonal) during and up to 6 months after trial therapy.

Subjects must satisfy all of the following additional criteria to be included in the OGT group:

1. No absolute contraindication for invasive procedures to obtain samples for organoid generation.
2. Sufficient material for organoid generation: biopsied samples (length>1cm, 2-3 pieces), surgically resected samples (>1cm×1cm×0.5cm, weight>200mg), malignant effusion samples collected by thoracentesis, abdominocentesis or lumbar puncture (pleural fluid>50mL, ascites>50mL, cerebrospinal fluid≥4 tubes with each tube ≥4mL).
3. Successful acquisition of a solid tumor biopsy sample containing ≥ 20% tumor content, or malignant effusion sample (e.g., pleural, or pericardial effusion or ascites) confirmed to contain malignant cells.

Exclusion Criteria:

1. Ineligible for all 5 of the study treatments either because of previously having received treatment in the advanced or metastatic setting or having a contraindication to treatment.
2. Documented mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious.
3. Known active central nervous system metastases, as indicated by clinical symptoms, cerebral edema, and/or progressive growth (patients with history of CNS metastases or spinal cord compression are eligible if they are clinically and radiologically stable for at least 4 weeks before first dose of trial treatment and have not required high-dose steroid treatment in the last 4 weeks).
4. Inflammatory breast cancer.
5. Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug product.
6. Major surgery within 3 weeks of starting study treatment: patients must have recovered from any effects of any major surgery.
7. Systemic treatment with anticancer therapy, antibody-based therapy, hormonal therapy, or radiotherapy within 3 weeks before study treatment.
8. Participation in a therapeutic clinical study within 3 weeks before study treatment, or current participation in other investigational procedures.
9. Has multiple primary malignancies within 3 years, except adequately resected nonmelanoma skin cancer, curatively treated in situ disease, or contralateral breast cancer.
10. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤1 or baseline.
11. Substance abuse or medical conditions such as clinically significant cardiac or pulmonary diseases or psychological conditions, that would, in the opinion of the Investigator, increase the safety risk to the subject or interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
12. Has known human immunodeficiency virus infection or active hepatitis B or C infection.
13. Has an uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.
14. Has gastrointestinal disorders likely to interfere with absorption of the study medication.
15. Is pregnant or breastfeeding or planning to become pregnant.
16. Any concurrent condition which in the Investigator's opinion makes it inappropriate for the patient to participate in the trial or which would jeopardize compliance with the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Through study completion, with an expected average of 1 year
  PFS is defined as the time from the date of randomization to the earliest date of the first objective documentation of radiographic disease progression according to RECIST version 1.1 or death due to any cause. Subjects who are alive with no objective documentation of (radiographic) disease progression by the data cutoff date for PFS analysis will be censored at the date of their last evaluable tumor assessment. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.

SECONDARY OUTCOMES:
Overall survival | Through study completion, with an expected average of 2 year
  OS is defined as the time from the date of randomization to the date of death for any cause. If there is no death reported for a subject before the data cutoff for OS analysis, OS will be censored at the last contact date at which the subject is known to be alive.
Objective response rate | Through study completion, with an expected average of 1 year
  ORR is defined as the sum of complete response (CR) rate and partial response (PR) rate according to RECIST version 1.1. CR is defined as disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR is defined as at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Disease control rate | Through study completion, with an expected average of 1 year
  DCR is defined as the sum of CR rate, PR rate, and stable disease (SD) rate. SD is defined as neither sufficient shrinkage to qualify for PR (taking as reference the sum of diameters at baseline) nor sufficient increase to qualify for PD (taking as reference the smallest sum of diameters while on study).
Clinical benefit rate | Through study completion, with an expected average of 1 year
  CBR is defined as the sum of CR rate, PR rate, and more than 6 months' SD rate.
Duration of response | Through study completion, with an expected average of 1 year
  DoR is defined as the time from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of disease progression, or death. DoR will be measured for responding subjects (PR or CR) only. Subjects who are progression-free at the time of the analyses will be censored at the date of the last evaluable tumor assessment.
Time to response | Through study completion, with an expected average of 1 year
  TTR is defined as the time from the date of randomization to the date of the first documentation of objective response (CR or PR). TTR will be measured for responding subjects (CR or PR) only.
Adverse events | Through study completion, with an expected average of 1 year
  Number of participants with adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China